CLINICAL TRIAL: NCT02199613
Title: Elvitegravir/Cobicistat/Tenofovir DF/Emtricitabine With Darunavir in Treatment-experienced Patients: Quality Control Monitoring of a Treatment Simplification Strategy
Brief Title: Elvitegravir/Cobicistat/Tenofovir DF/Emtricitabine With Darunavir Treatment Simplification Strategy
Acronym: QuaDar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Mark Hull, Clinical Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14-00490; H14-00490 (Other: UBC Providence Health Care Research Ethics Board)
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: HIV Infection
Keywords: HIV; antiretroviral therapy
MeSH Terms: conditions — HIV Infections | interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment simplification (Experimental): Open-label darunavir 800mg in conjunction with the co-formulated tenofovir DF/FTC/cobicistat/elvitegravir (Stribild) tablet, both taken together once daily with food
  Interventions: Drug: Treatment simplification

INTERVENTIONS:
Drug: Treatment simplification — Eligible, consenting subjects will start open-label darunavir 800mg plus the co-formulated tenofovir DF/FTC/cobicistat/elvitegravir (Stribild) tablet once daily with food, following the study procedures at the baseline visit. They will be assessed at weeks 2, 12, 24, 36, and 48 after starting the new regimen.
  Other Names: Darunavir 800mg plus Stribild tablet once daily

SUMMARY:
The study aims to assess the safety and efficacy of darunavir 800mg plus the co-formulated elvitegravir/cobicistat/tenofovir disoproxil fumarate (DF)/emtricitabine (Stribild) tablet as a simplification strategy for the treatment of HIV infection in HIV-infected subjects who have had previous antiretroviral treatment experience with multiple-drug regimens.

We hypothesize that elvitegravir/cobicistat/tenofovir DF/emtricitabine with darunavir will offer a safe and efficacious treatment simplification strategy for HIV positive patients currently receiving multiple-drug regimens to control their HIV infection.

DETAILED DESCRIPTION:
Eligible, consenting subjects will be assessed at baseline and weeks 2, 12, 24, 36, and 48. Study medications will be dispensed at all visits except week 2, and all participants will commence taking open-label darunavir 800mg in conjunction with the co-formulated tenofovir DF/emtricitabine/cobicistat/elvitegravir (Stribild) tablet, both taken together once daily with food, following study procedures at baseline.

Assessments at the study visits will include:

1. Complete physical exam including height and weight at baseline; symptom-directed physical exam and weight at other visits
2. Adverse clinical events including serious adverse events (hospitalizations etc.) and medication changes at every visit.
3. HIV RNA every 4 weeks.
4. CD4 and CD8 absolute counts and % at all visits except week 2.
5. Platelet count, aspartate amino transferase (AST), creatinine, estimated glomerular filtration rate (eGFR), phosphorus, urinalysis, and urine albumin to creatinine ratio (UACR) at each visit.
6. Fasting lipids (total, HDL, and LDL cholesterol and triglycerides), apolipoprotein B, high-sensitivity C- reactive protein (hsCRP) at baseline, week 24, and week 48.
7. Pregnancy test for women of child-bearing potential (as defined above) at every visit except week 2. In addition, pregnancy tests will be performed monthly for women of child-bearing potential; between study visits these may be done at home.
8. A plasma sample (3 mL) will be collected and stored once at baseline for all subjects, and used for measurement of darunavir trough (pre-dose) concentration in subjects receiving darunavir in their pre-study regimen.
9. All subjects will take their study medication under observation in the clinic on Day 14, and plasma samples (3mL) for pharmacokinetic testing will be drawn immediately pre-dose and at 1, 2, 3, 4, 5, 6, and 8 hours post-dose. Subjects will return the following day before taking their Day 15 dose for a 24-hour post-dose sample.
10. Peripheral blood mononuclear cells (PBMCs) will be collected and stored at baseline for possible future study-related testing.
11. The following questionnaires will be completed by participants prior to other study procedures at baseline and at weeks 24 and 48: MOS-HIV quality of life questionnaire; HIVTSQ; ACTG treatment adherence questionnaire; and the medication adherence self-report inventory (MASRI).

ELIGIBILITY:
Inclusion Criteria:

* HIV positive adults > or = 19 years of age
* receiving stable therapy including one or two nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs), in conjunction with a once-daily protease inhibitor (PI) (atazanavir, lopinavir or darunavir) and twice daily raltegravir or once daily dolutegravir
* Virologic suppression for >6 months, defined as plasma viral load (VL) consistently < 200 copies/mL with no evidence of prior virologic rebound (VL > 1000 copies/mL) on the NRTI/PI/Raltegravir regimen, AND VL < 50 copies/mL at time of study screening
* Estimated glomerular filtration rate (eGFR) > o r= 70mL/min at screening

Exclusion Criteria:

* Prior documented viral rebound > 1000 copies/mL on any raltegravir-containing regimen
* Evidence of resistance mutations compromising raltegravir or elvitegravir activity on prior genotypes.
* Evidence of clinically significant resistance to tenofovir on any previous genotype tests: K65R mutation, or 3 or more thymidine-analogue associated mutations (TAMS) compromising tenofovir activity
* Evidence of resistance mutations significantly compromising darunavir activity on any previous genotypic tests
* Current use of any nonnucleoside reverse transcriptase inhibitor (NNRTI)
* Pregnancy or breast-feeding
* Contraindications to tenofovir/FTC, elvitegravir, or cobicistat (e.g. previous significant toxicity, intolerance or drug interactions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Plasma HIV RNA | 12 weeks
  Proportion of individuals with plasma HIV RNA <200copies/mL at 12 weeks following regimen switch

SECONDARY OUTCOMES:
plasma HIV RNA | weeks 12, 24 and 48
  Proportion of individuals with plasma HIV RNA < 50 copies/mL at weeks 12, 24 and 48 post switch
plasma HIV RNA | week 24 and 48
  Proportion of individuals with plasma HIV RNA < 200 copies/mL at week 24 and 48 post switch
CD4 cell count, CD4% and CD4/CD8 ratio | 12, 24 and 48 weeks
  Change in CD4 cell count, CD4% and CD4/CD8 ratio from study baseline to 12, 24 and 48 weeks after switch.
serum creatinine and estimated glomerular filtration rate (eGFR) | 12, 24, and 48 weeks
  Change in serum creatinine and eGFR from baseline to 12, 24 weeks and 48 weeks.
Adverse event discontinuations | 48 weeks
  Proportion of adverse events experienced necessitating switch to original regimen
fasting lipid parameters (total cholesterol, LDL, HDL, triglycerides, and apolipoprotein B [apoB]), AST to platelet ratio index (APRI) score, and high-sensitivity C-reactive protein (hsCRP) | 24 and 48 weeks
  Changes in fasting lipid parameters (total cholesterol, LDL, HDL, triglycerides, and apolipoprotein B [apoB]), AST to platelet ratio index (APRI) score, and high-sensitivity C-reactive protein (hsCRP) between baseline and 24 and 48 weeks.
Darunavir plasma concentration | week 2
  Change in darunavir trough concentration from baseline to week 2 for individuals receiving darunavir at baseline
HIV Treatment Satisfaction Questionnaire (HIVTSQ) scores and quality of life indicators (MOS-HIV scores) | weeks 24 and 48
  Changes in HIV Treatment Satisfaction Questionnaire (HIVTSQ) scores and quality of life indicators (MOS-HIV scores) between baseline and weeks 24 and 48 following switch.
Adherence | 24 and 48 weeks
  Changes in antiretroviral adherence from baseline to 24 and 48 weeks. Adherence will be assessed using two measures: the ACTG treatment adherence questionnaire and the Medication adherence self-report inventory (MASRI).
Elvitegravir plasma concentrations | Day 14
  Elvitegravir concentrations will be measured at day 14
Adverse events | 48 weeks
  Adverse events necessitating a resumption of the previous antiretroviral regimen, and all serious adverse events will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hull, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital Immunodeficiency Clinic, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Harris M, Ganase B, Watson B, Harrigan PR, Montaner JSG, Hull MW. HIV treatment simplification to elvitegravir/cobicistat/emtricitabine/tenofovir disproxil fumarate (E/C/F/TDF) plus darunavir: a pharmacokinetic study. AIDS Res Ther. 2017 Nov 2;14(1):59. doi: 10.1186/s12981-017-0185-4. PMID 29096670